CLINICAL TRIAL: NCT06047171
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Intravenously Administered ALE.F02 to Evaluate the Safety, Tolerability, Pharmacokinetics, and Renal Sparing in Antineutrophil Cytoplasmic Antibody-Associated Vasculitis With Rapidly Progressive Glomerulonephritis
Brief Title: Rescue of Nephrons With ALE.F02 (RENAL-F02)
Acronym: RENAL-F02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alentis Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALE.F02.03; 2022-502184-38 (Other: EU Clinical Trial Number); U1111-1286-9095 (Other: WHO universal trial number (UTN))
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Glomerulonephritis Rapidly Progressive
MeSH Terms: interventions — Rituximab; Glucocorticoids; Cyclophosphamide; Immunosuppressive Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard treatment + ALE.F02 low dose infusions (Experimental): Standard treatment + ALE.F02 low dose infusions
  Interventions: Biological: ALE.F02; Drug: Rituximab; Drug: GlucoCorticoid; Drug: Cyclophosphamid; Drug: Immunosuppressive Agents
- Standard treatment + ALE.F02 high dose infusions (Experimental): Standard treatment + ALE.F02 high dose infusions
  Interventions: Biological: ALE.F02; Drug: Rituximab; Drug: GlucoCorticoid; Drug: Cyclophosphamid; Drug: Immunosuppressive Agents
- Standard treatment + placebo infusions (inactive substance) (Placebo Comparator): Standard treatment + placebo infusions (inactive substance)
  Interventions: Drug: Rituximab; Drug: GlucoCorticoid; Drug: Cyclophosphamid; Drug: Placebo; Drug: Immunosuppressive Agents
- Standard treatment + ALE.F02 maximum dose infusions (Experimental): Standard treatment + ALE.F02 maximum dose infusions
  Interventions: Biological: ALE.F02; Drug: Rituximab; Drug: GlucoCorticoid; Drug: Cyclophosphamid; Drug: Immunosuppressive Agents

INTERVENTIONS:
Biological: ALE.F02 — ALE.F02 is an anti-Claudin-1 (CLDN1) monoclonal antibody (mAb) to selectively target the non-tight junctions (TJ), exposed form of CLDN1. CLDN1 is an integral component of the TJs between cells.
  Arms: Standard treatment + ALE.F02 high dose infusions; Standard treatment + ALE.F02 low dose infusions; Standard treatment + ALE.F02 maximum dose infusions
Drug: Rituximab — Rituximab is a monoclonal antibody that targets cluster of differentiation antigen 20 (CD20), an antigen expressed on the surface of pre-B and mature B-lymphocytes
Drug: GlucoCorticoid — Glucocorticoids are a class of corticosteroids, which are a class of steroid hormones that bind to the glucocorticoid receptor. Glucocorticoid effects may be broadly classified into two major categories: immunological and metabolic.
Drug: Cyclophosphamid — Cyclophosphamid is a medication used as chemotherapy and to suppress the immune system
Drug: Placebo — Drug product that will contain no active ingredient
  Arms: Standard treatment + placebo infusions (inactive substance)
Drug: Immunosuppressive Agents — Immunosuppressants are drugs that prevent your immune system from attacking healthy cells and tissues by mistake.

SUMMARY:
The goal of this clinical trial is to learn if a new drug that might help protect and preserve kidney function in antineutrophil cytoplasmic antibody (ANCA) associated vasculitis (AAV). AAV is a type of autoimmune disease where the body's own immune system attacks itself, and in the case of AAV the body attacks its own small blood vessels. There are many small blood vessels in the kidneys meaning the kidneys are commonly affected in AAV.

The main questions it aims to answer are:

* Is the new drug well tolerated and safe?
* Can the new drug protect and preserve kidney functions when is added to standard therapy?

Researchers will compare the following groups to see how the new drug is tolerated and what effect to preserve kidney tissue has:

* Group A: Standard treatment + ALE.F02 low dose infusions
* Group B: Standard treatment + ALE.F02 high dose infusions
* Group C: Standard treatment + ALE.F02 maximum dose infusions
* Group D: Standard treatment + placebo infusions (inactive substance)

The Treatment period will consist of 24 weeks beginning on Day 1, during which time participants will receive 13 infusions of the study medicine, along with standard therapy for kidney inflammation due to AAV. During the treatment period, participants will have the following assessments:

* A brief physical examination focusing on their skin any pre-existing medical conditions that you have.
* Collection of blood and urine samples for routine safety tests and to assess renal function.
* Collection of blood samples:

  * To measure the amount of study medicine in their blood. This is called pharmacokinetics (PK) and it is tested to see how study medicine enters, moves through, and exits the body.
  * To test for antidrug antibodies (ADA). To check if their body create antibodies against the study medicine, as this could reduce its effect.
  * To measure biomarkers. Biomarkers are specific compounds in the body (can be protein, hormones, or genetic molecules) that indicate normal or abnormal processes taking place in your body and may be a sign of an underlying condition or disease (for example glucose levels are used as biomarker in managing diabetes). They are used to see how well the body responds to a treatment for a disease or condition.
* Collection of urine to measure urine markers of vasculitis/inflammation called biomarkers.
* Urine pregnancy test. A urine pregnancy test is a quick medical test that can tell if a woman is pregnant or not by checking for a hormone which is produced during pregnancy, usually in the urine.
* Chest High Resolution Computed Tomography (HRCT) scan to check whether they have vasculitis affecting their lungs. A CT scan uses special x-ray equipment to take detailed pictures of body tissues and organs to diagnose and monitor conditions in various parts of the body. For the CT scan, they will need to lie still on a table. At Week 24 a second lung CT scan will be performed for participants whose initial scan showed lung vasculitis to see whether your lung vasculitis is getting better or ongoing/worse.

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female patients ≥18 years of age of any race or ethnicity with a score of <7 on the Clinical Frailty Scale in the 3 months preceding the onset of RPGN attributed to AAV; Note: The PI should assess the Clinical Frailty Scale based on medical history and interview with the patient
2. Must be willing and able to comply with the study requirements and give informed consent for participation in the study;
3. Must be willing to have a renal biopsy procedure performed no later than prior to study drug administration at the Week 6 Visit; alternatively, a historical biopsy performed up to 45 days prior to the initiation of study drug administration is considered acceptable;
4. Have been newly diagnosed with RPGN within 45 days prior to the initiation of study drug treatment, as demonstrated by the following: - Evidence of loss of renal function with an eGFR of ≤50 mL/min/1.73 m2 and ≥10 mL/min/1.73 m2; and - History of proteinuria of any degree AND/OR hematuria that is temporally associated with the presenting episode of illness and supports the diagnosis of RPGN. Note: The hematuria may be represented by the presence of eumorphic or dysmorphic red blood cells (RBCs) and/or RBC casts. Patients with extrarenal manifestations of ANCA which started prior to RPGN should be discussed with the Medical Monitor and the Sponsor.
5. Are suspected of having RPGN attributed to AAV at Screening based on clinical laboratory diagnostic criteria, including a positive test for an ANCA, ie, anti-myeloperoxidase (MPO) or anti-proteinase 3 (PR3);
6. Have a body weight of ≤130 kg;
7. Female patients must not be pregnant or lactating at Screening and 1 of the following conditions must apply: - Is a female of childbearing potential and agrees to use a highly effective method of birth control during their participation in the study and for at least 5 half-lives or a minimum of 30 days after the last dose of study drug, or as recommended in the Summary of Product Characteristics (SmPC) of any authorized AxMP given as part of background standard of care (SOC) therapy, whichever is longer; or - Is a female of nonchildbearing potential.
8. Female patients must agree not to donate ova for 6 months after the last dose of study drug or as recommended in the SmPC of any authorized AxMP given as part of background SOC therapy, whichever is longer;
9. Male patients must agree to use contraception, in the form of either sexual abstinence or a condom, during their participation in the study and for 90 days after the last dose of study drug or as recommended in the SmPC of any authorized auxiliary medicinal product (AxMP) given as part of background SOC therapy, whichever is longer; and
10. Male patients must agree to abstain from sperm donation during their participation in the study and for 90 days after the last dose of study drug or as recommended in the SmPC of any authorized AxMP given as part of background SOC therapy, whichever is longer.

Exclusion Criteria:

1. Have a history of previous RPGN that resolved or ameliorated (ie, the patient had a documented case of RPGN and has suffered a relapse);
2. Have a positive serology test for anti-glomerular basement membrane antibodies;
3. Have evidence of active or latent tuberculosis (TB) determined by a positive (not indeterminate) QuantiFERON®-TB Gold test (or equivalent). In countries where QuantiFERON®-TB Gold test (or equivalent) is not available, radiological criteria, including chest X-ray or computed tomography scan, may alternatively be used;
4. Have a chronic infection that could be exacerbated by RPGN or SOC therapy for RPGN;
5. Have active hepatitis B, hepatitis C, or HIV infection;
6. Have taken any prohibited medications.
7. Have received a course of SOC therapy which exceeds a high-dose prolonged regimen of treatment of ANCA RPGN, such as >3000 mg of IV methylprednisolone-equipotent glucocorticoids, or >1 mg/kg/day of oral glucocorticoids (prednisone equivalent) for >14 days (doses are provided as a guidance for assessment of intensity; patients who received high-dose glucocorticoids should be discussed with and approved by the Medical Monitor and the Sponsor); Note: A course of systemic glucocorticoids attributed to extrarenal manifestation of ANCA should not be included in the assessment of Exclusion Criterion 7 and such occasions should be discussed with the Medical Monitor and the Sponsor. IV methylprednisolone administered as pre-medication for rituximab may be considered as prophylaxis of a potential hypersensitive response to rituximab. This pre-medication is allowed during the course of the study and will not account in the total dose calculation of the IV glucocorticoids threshold of 3000 mg at Screening for eligibility assessment.
8. Have been treated or planned to be treated with avacopan;
9. Have poor venous access;
10. Have participated in an investigational drug or device study and received investigational therapy <30 days or 5 half lives, whichever is the greater, prior to the first dose of study drug. For biological investigational drugs, the exclusionary period may not be <90 days prior to the first dose of study drug;
11. Have a history of psoriasis, AD, excessively dry skin or recurrent conjunctivitis that has required treatment prescribed by a physician, scleroderma, vitiligo, or any other active autoimmune dermatological disorder, with the exception of dermatological disorders or skin rashes that are attributable to, or known to be associated with, the underlying diagnosis of AAV, which shall not be exclusionary;
12. Have a diagnosis of systemic lupus erythematosus-AAV overlap syndrome;
13. Have a diagnosis of eosinophilic granulomatosis with polyangiitis;
14. Have evidence of uncontrolled respiratory, cardiac, hepatic, endocrine, central nervous system, or renal disease, unrelated to RPGN or AAV, that the PI believes cannot be readily brought under control, or any other medical condition that in the opinion of the PI renders the patient unsuitable for enrollment and could prevent the successful completion of the study;
15. Have received a live vaccine within 30 days prior to Screening;
16. Have received any vaccine within 7 days of the first dose of study drug other than against influenza or pneumococcal infection;
17. Are employed by the PI or the study site, have direct involvement in the proposed study or other studies under the direction of that PI, or are a family member of the PI or study site personnel;
18. Have not recovered from AEs and/or complications from major surgery prior to the first dose of study drug; Note: The PI should consult with the Medical Monitor and Sponsor to determine if ongoing, significant complications from major surgery are exclusionary.
19. Have active or known history of alcohol or substance abuse within 1 year prior to Day 1/Randomization or have a positive urine drug screen for drugs of abuse at Screening;
20. Have been diagnosed within the preceding 5 years with a malignant neoplastic disease, other than locally invasive cutaneous squamous or basal cell carcinoma;
21. Have alveolar haemorrhage with hypoxia defined by an oxygen saturation <85% or that requires the use of invasive or noninvasive ventilatory support;
22. Have undergone dialysis within 7 days prior to Screening;
23. Have undergone therapeutic plasma exchange within 7 days prior to the first dose of study drug; or
24. Have known hypersensitivity to the study drug or any of the excipients used in the formulation of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint for this study is the safety and tolerability of ALE.F02 when administered as a continuous IV infusion in patients with rapidly progressive glomerulonephritis (RPGN) attributed to AAV. | through study completion, an average of 1 year
  Safety endpoints are the following:
  * All adverse events (AEs);
  * All serious adverse events (SAEs);
  * Hematology and clinical chemistry analyte assessments;
  * Serum lipids;
  * Antidrug antibodies (ADAs); and
  * ECGs

SECONDARY OUTCOMES:
The key secondary endpoint for this study is the change in mean estimated glomerular filtration rate (eGFR) from baseline to Week 24/End of Treatment (EOT) for recipients of ALE.F02 compared to placebo. | from baseline to Week 24/EOT
Change in mean urine protein to creatinine ratio (UPCR) area under the concentration time curve (AUC) from baseline to Week 24/EOT for recipients of ALE.F02 compared to placebo; | from baseline to Week 24/EOT
Change in mean urine protein to creatinine ratio (UPCR) area under the concentration time curve (AUC) from baseline to Week 52/End of Study (EOS) for recipients of ALE.F02 compared to placebo; | from baseline to Week 52/EOS
Time to stable proteinuria (≤0.5 g/day for ≥14 days) during the Treatment Period for recipients of ALE.F02 compared to placebo; | up to 24 weeks
Time to stable hematuria (≤5 RBCs/high-power field for ≥14 days) during the Treatment Period for recipients of ALE.F02 compared to placebo; | up to 24 weeks
Incidence of renal replacement therapy (RRT) at any time during the study for recipients of ALE.F02 compared to placebo; and | through study completion, an average of 1 year
Total glucocorticoid and immunosuppressive exposure at Week 24/EOT and Week 52/EOS for recipients of ALE.F02 compared to placebo. | at Week 24/EOT and Week 52/EOS

CONTACTS AND LOCATIONS:
Locations (49):
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- France (10):
  - Centre Hospitalier Boulogne sur Mer, Boulogne-sur-Mer, Cedex
  - CHU Bordeaux - Hopital Pellegrin, Bordeaux
  - CHRU de Brest - Hopital de la Cavale Blanche, Brest
  - CHU Grenoble-Alpes - Hopital Michallon, La Tronche
  - CHU de Nantes - Hotel-Dieu, Nantes
  - CHU de Nimes, Nîmes
  - AP-HP Hopital Pitie-Salpetriere, Paris
  - AP-HP Hopital Cochin, Paris
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - Centre Hospitalier de Valenciennes, Valenciennes
- Germany (8):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Koeln (AoeR), Cologne
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München
- Italy (5):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
  - APSS Ospedale Santa Chiara di Trento, Trento
- Spain (5):
  - Fundacio Puigvert, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
- Sweden (2):
  - Linkoping University Hospital, Linköping
  - University Hospital of Umea, Umeå
- Switzerland (4):
  - Kantonsspital Baden AG, Baden
  - Inselspital, Universitaetsspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - Hôpital Fribourgeois-Freiburger Spital, Villars-sur-Glâne
- Turkey (Türkiye) (4):
  - Ankara Etlik City Hospital, Ankara, Keçiören
  - Marmara University Medical Faculty Hospital, Istanbul
  - Kocaeli University Medical School - Internal Medicine - Nephrology, Kocaeli
  - Erciyes University Faculty of Medicine, Melikgazi
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Cambridge University - Addenbrooke's Hospital, Cambridge
  - Royal Liverpool University Hospital, Liverpool
  - Imperial College Healthcare NHS Trust, London
  - Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: Undecided